CLINICAL TRIAL: NCT02919527
Title: Acute Effects of Foam Rolling on Viscoelastic Tissue Properties and Fascial Sliding: A Randomized, Controlled Crossover Trial
Brief Title: Acute Effects of Foam Rolling on Viscoelastic Tissue Properties and Fascial Sliding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dr. Winfried Banzer, Head of Department, Goethe University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SpM2016-005
Record Dates: First submitted 2016-09-27; First posted 2016-09-29 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Fascia; Self-Myofascial-Release; Passive Stiffness; Fascial Sliding; Flexibility

ARMS (3):
- Self-Myofascial-Release (Experimental): Two 60 seconds bouts of Self-Myofascial-Release performed at the anterior thigh; anticipated intensity of 7/10 on a 10 point numeric rating scale (0 representing no discomfort and 10 representing maximal discomfort)
  Interventions: Other: Self-Myofascial-Release
- Stretching (Active Comparator): Two 60 seconds bouts of static stretching performed at the anterior thigh; anticipated intensity of 7/10 on a 10 point numeric rating scale (0 representing no discomfort and 10 representing maximal discomfort)
  Interventions: Other: Stretching
- Control (No Intervention): No Intervention

INTERVENTIONS:
Other: Self-Myofascial-Release — Self-Myofascial-Release performed at the anterior thigh
  Arms: Self-Myofascial-Release
Other: Stretching — Static Stretching performed at the anterior thigh
  Arms: Stretching

SUMMARY:
Treatment or training of fascial tissues has moved into the focus of medical research in the last decade. In this context, the use of foam rollers or roller massagers for self-myofascial-release (SMR) techniques has become increasingly popular in health and fitness professionals. The primary objective of these techniques is to mimic manual massage or myofascial-release therapy with a self-usable tool. Recent studies suggest that SMR improves, inter alia, range of motion (ROM) without a decrease in neuromuscular performance (Cheatham et al. 2015).

Concurrent effects on the muscle and especially the surrounding connective tissue network have been proposed as underlying mechanisms for these observed changes in ROM after SMR. Several authors assume a positive effect of SMR on sliding properties of different independent fascial layers. Also, changes in passive tissue stiffness is suggested. Passive stiffness is thereby characterized by passive resistance in the tissues' (muscles') functional direction, the passive resistive torque (PRT).

In conclusion, for many of the proclaimed effects of SMR, such as improvements of sliding of fascial layers or decreases of passive stiffness, there is a lack of evidence in the literature. Therefore, the aim of the study is to evaluate acute effects of SMR on the viscoelastic properties of the muscles on the anterior thigh and the corresponding fascia.

In a cross over design, 16 subjects receive all of the following interventions after a familiarization session: a) 2x60 seconds of SMR at the anterior thigh, b) 2x60 seconds of static stretching at the anterior thigh, c) no intervention in a balanced permutated randomization sequence. Before and directly after each intervention, outcome parameters are collected.

Passive Resistive Torque is evaluated using a computerized isokinetic dynamometer. In passive mode, the lower leg is moved from full knee extension (0°) to the point of maximal knee flexion with a velocity of 5°/s. Torque and angle are recorded at 100 Hertz (Hz). Sliding of fascial layers is quantified with a frame-by-frame cross correlation algorithm of high-resolution ultrasound images (Dilley et al. 2001).

First stretch sensation is quantified using the passive mode in the isokinetic dynamometer.

Maximal ROM is detected using a an ultrasonographic movement analysis system in a prone position.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-40 years

Exclusion Criteria:

* History of orthopedic injuries in the lower extremity in the last 12 months
* Any history of psychiatric, cardiovascular, endocrine, neurological, or metabolic disorders
* Any current medication that might affect pain perception or proprioception
* Muscle soreness
* Pregnancy/nursing period
* Nonspecific musculoskeletal disorders

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-09; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Passive-Resistive-Torque, Biodex System 3 Professional | 1 minute
  In passive mode, the lower leg is moved from full knee extension (0°) to the point of maximal knee flexion with a velocity of 5°/s. Torque and angle are recorded at 100 Hz, and passive stiffness can be calculated from the torque-angle relationship.
Fascial-Sliding, Siemens Acuson X300, Cross correlation | 1 minute
  Sliding of fascial layers is quantified with a frame-by-frame cross correlation algorithm of high-resolution ultrasound images. The cross-correlation method calculates the correlation coefficient between the pixel grey levels for selected rectangle-shaped regions of interest (ROIs) in two adjacent images. The pixel shift that gives the maximum correlation coefficient corresponds to the relative movement between two frames.

SECONDARY OUTCOMES:
Maximal Range of Motion, Zebris CMS20 | 1 minute
  A triplet of ultrasonographic markers is placed on the lower leg, a second triplet is placed as a reference on the thigh. Participants are placed on a physio table including a pre-stretch of the hip (210° in total) using a bed wedge (30°). In this position, participants are instructed to perform three consecutive active knee flexion-extension cycles at a self-selected velocity. Subsequently, the investigator performs three passive knee flexion-extension cycles. Movements are recorded in three dimensions at 20 Hz, and maximal active as well as passive ROM can be calculated as the maximal displacement relative to the starting position recorded by the US markers.
First stretch sensation, Biodex System 3 Professional | 1 minute
  Position of the first stretch sensation is quantified using the isokinetic dynamometer in the above-described position. In passive mode, the knee is flexed from full extension to flexion at 5°/s. The subject uses a switch to stop the passive movement at the position of first stretch sensation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sports Medicine, Goethe University Frankfurt/Main, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Cheatham SW, Kolber MJ, Cain M, Lee M. THE EFFECTS OF SELF-MYOFASCIAL RELEASE USING A FOAM ROLL OR ROLLER MASSAGER ON JOINT RANGE OF MOTION, MUSCLE RECOVERY, AND PERFORMANCE: A SYSTEMATIC REVIEW. Int J Sports Phys Ther. 2015 Nov;10(6):827-38. PMID 26618062
- [Background] Dilley A, Greening J, Lynn B, Leary R, Morris V. The use of cross-correlation analysis between high-frequency ultrasound images to measure longitudinal median nerve movement. Ultrasound Med Biol. 2001 Sep;27(9):1211-8. doi: 10.1016/s0301-5629(01)00413-6. PMID 11597362
- [Derived] Krause F, Wilke J, Niederer D, Vogt L, Banzer W. Acute effects of foam rolling on passive tissue stiffness and fascial sliding: study protocol for a randomized controlled trial. Trials. 2017 Mar 9;18(1):114. doi: 10.1186/s13063-017-1866-y. PMID 28274273